CLINICAL TRIAL: NCT04729595
Title: A Phase 2/3, Adaptive, Randomized, Double-Blind, Placebo-Controlled Study to Examine the Effects of Tempol (MBM-02) in Subjects With COVID-19 Infection
Brief Title: Study to Evaluate the Effects of Tempol (MBM-02) in COVID-19 Patients.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study did not demonstrate statistical significance of its primary endpoint of clinical resolution of COVID-19 symptoms at day 14 versus placebo
Sponsor: Adamis Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC400-03
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — tempol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, placebo-controlled enrolling high risk subjects with early COVID19 infection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, Double-blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): Tempol (MMB-02) 800 mg per Day (n=124)
  Interventions: Drug: Tempol
- Placebo (Placebo Comparator): Placebo (n=124)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tempol — Tempol 800 mg capsule will be administered at 400mg (2 capsules) two times daily for fourteen (14) consecutive days.
  Arms: Active Treatment
Other: Placebo — Placebo capsules will be administered orally (2 capsules) two times daily for fourteen (14) consecutive days.
  Arms: Placebo

SUMMARY:
An Adaptive, Randomized, Double-blind, Placebo-controlled study to examine the Effects of Tempol in subjects with COVID-19 infection.

DETAILED DESCRIPTION:
Phase 2/3 Adaptive, Randomized, Double-blind, placebo-controlled enrolling high risk subjects with early COVID19 infection with a primary endpoint of limiting hospitalization.

As part of the initial phase 2 portion of the study, 50 COVID positive subjects with comorbidities will be enrolled. Eligible subjects positively diagnosed COVID-19 infection will be randomized 1:1 to receive either Tempol or placebo.

An interim analysis by a DSMB will examine safety and markers of systemic inflammation during a Stage 1 interim analysis. Based on the DSMB adjudication, the Phase 3 portion of the trial will begin with a second interim analysis after enrollment of 124 subjects

This protocol will seek to enroll approximately 248 subjects > 18 years of age diagnosed with COVID-19 infection. All subjects will receive standard of care. As standard of care can vary between institution over time for the treatment of COVID-19; Off label medication use, therapies, devices, and interventions used in standard of care practice for COVID-19 is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and above with at least one risk factor for disease progression (i.e., age≥ 65, hypertension, diabetes, obesity (BMI ≥30 as defined by CDC), cancer, immunodeficiency and in the opinion of the investigator the risk factor is not acutely life-threatening).
* Laboratory confirmed infection of SARS-CoV-2 within 5 days of Baseline/day 1.
* Subjects must meet the severity score of Moderate or greater for two of the first ten symptoms listed in the Patient Reported Outcomes (PRO) at screening.
* Ability to travel to clinic.
* Ability to understand and sign an informed consent form.
* Female subjects of child-bearing potential who are capable of conception must be: post- menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing two effective methods of birth control. Acceptable methods include abstinence, intrauterine device, spermicide, barrier, male partner surgical sterilization and hormonal contraception. A female subject ≥18 years of age and of child bearing potential must agree to practice two acceptable methods of birth control during the study period.
* Ability to swallow a capsule.
* Ability to complete an electronic diary via smartphone or web.

Exclusion Criteria:

* Need for hospitalization based on severe or critical symptoms based on CDC guidance.
* Subject in long-term care facility.
* Known hypersensitivity or contra-indication to Tempol.
* Subjects taking STRONG CYP inhibitors (e.g. fluoxetine, itraconazole, quinidine, clarithromycin).
* In the opinion of the investigator, any reason that would make the follow up of the subject impossible during the study treatment and follow up period. Any reason the subject cannot comply with study and study procedures.
* Subjects receiving any other investigational agent within 4 weeks of Baseline/Day 1.
* Use of non-FDA approved (EUA or full approval)/off label treatments for COVID-19.
* Lactating females.
* History of any known chronic liver or kidney disease.
* Subjects taking drugs with a Narrow Therapeutic Index such as Cyclosporine Digoxin Flecainide Lithium Phenytoin Sirolimus Theophylline, and Warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of sustained clinical resolution1 of symptoms of COVID-19 | 14 Days from the date Randomization/First Dosing.
  To evaluate the difference in the rate of sustained clinical resolution1 of symptoms of COVID-19 at Day 14 by evaluating the odds ratio of the rate of sustained clinical resolution1 of symptoms of COVID-19 between Tempol + SOC vs placebo + SOC at Day 14.

SECONDARY OUTCOMES:
Safety of Tempol + SOC vs placebo + SOC: Occurrence of Adverse Events/All cause of mortality | 60 Days from Randomization/First Dosing.
  To evaluate the safety of Tempol + SOC vs placebo + SOC from Baseline/Day 1 through Day 60 For:
  * Occurrence of treatment-emergent adverse events (TEAEs).
  * Occurrence of TEAEs leading to withdrawal of study treatment or premature study discontinuation.
  * All cause of mortality (death of the patient, from any cause).
Efficacy of Tempol on preventing hospitalization: Odds ratio of the rate of hospitalization | 14 Days from the date Randomization/First Dosing.
  To evaluate the efficacy of Tempol on preventing hospitalization at Day 14 in subjects with COVID-19 by evaluating the odds ratio of the rate of hospitalization in subjects with COVID-at Day 14 between treatment arms.
Changes in functional status: Post COVID Functional Scale (PCFS) | 7,14 and 21 Days from the date Randomization/First Dosing.
  To evaluate the changes in functional status measured by Post COVID Functional Scale (PCFS) at Baseline/Day1 to Day7, Day 14 and Day 21 by evaluating the difference in the Post COVID Functional Scale (PCFS) measurement between Tempol + SOC vs. placebo + SOC. The scale is measured from 0 - 10, with a higher score being worse.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Moss, MD, Study Director — Adamis Pharmaceutical Corporation
Locations (17):
- United States (17):
  - Pinnacle Research Group, Anniston, Alabama
  - LA Universal Research, Los Angeles, California
  - Doral medical Research, Doral, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Center for Respiratory and Sleep Medicine, Greenwood, Indiana
  - Tandem Clinical Research GI, LLC., Marrero, Louisiana
  - Barrett Clinical, La Vista, Nebraska
  - Monroe Biomedical Research, Monroe, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - Vilo Research Group, Houston, Texas
  - United Memorial Medical Center, Houston, Texas
  - R&H Clinical Research, Katy, Texas
  - Meridian Clinical Research, Portsmouth, Virginia
  - Eastside Research Associates, Redmond, Washington

IPD SHARING:
Plan to Share IPD: Undecided